CLINICAL TRIAL: NCT06466681
Title: Changes in Attentional Control After a Focal Seizure.
Acronym: ATTENTIONEPIF
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2022_0762
Record Dates: First submitted 2024-05-21; First posted 2024-06-20 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Temporal Lobe Epilepsy; Frontal Lobe Epilepsy; Others Subtypes
Keywords: Attentional control; Focal epilepsy; Event related potentials; Functionnal connectivity; high-resolution EEG
MeSH Terms: conditions — Epilepsy, Temporal Lobe; Epilepsy, Frontal Lobe; Epilepsies, Partial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: All included subjects — Administration of the subtest of divided attention of the Test of Attentional Performance (TAP), recording of the event related potentiels N200 and P300, measure of the variation of power in several frequency bands (theta, alpha and beta) and measure of the high-resolution EEG connectivity during an attentional task at several time-points : a first time during interictal period (no seizure for more than 24 hours) and 1, 3, 6 and 24 hours after a focal seizure.

SUMMARY:
Epilepsy is frequently associated with cognitive and attentional disorders. Several studies have pointed out that there are modifications of brain activity in resting state during peri-ictal period in EEG and functional MRI. However, to date, no study has assessed the changes in attentional control after a seizure. The investigators hypothesize that a localized discharge is associated with a disorganization of the networks engaged in attentional control. In this regard, the investigators propose a prospective longitudinal study assessing the changes in attentional control after a focal seizure.

ELIGIBILITY:
Inclusion Criteria:

* Age superior to 18 and under 80
* Focal epilepsy with indication to pre-surgery work-up and 5 days programmed hospitalization dedicated to this work-up
* Normal global cognitive performance (standard progressive Raven matrices score > 5th percentile)
* Be affiliated to the social security system
* Have signed an informed consent

Exclusion Criteria:

* Pregnancy or breastfeeding
* Not able to give consent (Article 1121-8 of the CSP)
* Vulnerable person
* Being deprived of liberty by judicial or administrative decision (Article L 1121-6 of the CSP)
* Guardianship
* Have a high probability of not respecting the protocol or of abandoning the study
* Absence of any epileptic seizure recorded during the hospitalization
* Recurrent seizures preventing the recording of at least 24 hours without any seizure following a seizure.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Administration of the subtest of divided attention of the Test of Attentional Performance (TAP), recording of the event related potentiels N200 and P300, measure of the variation of power in several frequency bands (theta, alpha and beta) and measure of the high-resolution EEG connectivity during an attentional task at several time-points : a first time during interictal period (no seizure for more than 24 hours) and 1, 3, 6 and 24 hours after a focal seizure.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-03-04 (Actual); Primary Completion 2027-03-09 (Estimated); Study Completion 2027-03-09 (Estimated)

PRIMARY OUTCOMES:
Subtest of divided attention of the Test of Attentional Performance (TAP) | 24 hours
  A first time during interictal period (no seizure for more than 24 hours) (this first measure will be repeated every day until a seizure is recorded) and 1, 3, 6 and 24 hours after a focal seizure.

SECONDARY OUTCOMES:
N200 amplitude and latency | 24 hours
  A first time during interictal period (no seizure for more than 24 hours) (this first measure will be repeated every days until a seizure is recorded) and 1, 3, 6 and 24 hours after a focal seizure.
Strength of EEG functionnal connectivity during an attentional task (global and regional) | 24 hours
  A first time during interictal period (no seizure for more than 24 hours) (this first measure will be repeated every days until a seizure is recorded) and 1, 3, 6 and 24 hours after a focal seizure.
Variation of power in several frequency bands (theta, alpha and beta) during an attentional task. | 24 hours
  A first time during interictal period (no seizure for more than 24 hours) (this first measure will be repeated every day until a seizure is recorded) and 1, 3, 6 and 24 hours after a focal seizure.
Magnetic resonance imaging functional connectivity. | up to 5 days
Differences in N200 and P300 amplitude and latency recorded between different subgroups according to the epileptic focus. | 24 hours
  A first time during interictal period (no seizure for more than 24 hours) (this first measure will be repeated every day until a seizure is recorded) and 1, 3, 6 and 24 hours after a focal seizure.
P300 amplitude and latency | 24 hours
  A first time during interictal period (no seizure for more than 24 hours) (this first measure will be repeated every days until a seizure is recorded) and 1, 3, 6 and 24 hours after a focal seizure.
Differences in strength of EEG functional connectivity during an attentional task recorded between different subgroups according to the epileptic focus. | 24 hours
Differences in variation of power in several frequency bands (theta, alpha and beta) during an attentional task recorded between different subgroups according to the epileptic focus. | 24 hours
Differences in magnetic resonance imaging functional connectivity recorded between different subgroups according to the epileptic focus. | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital,, Lille, France

IPD SHARING:
Plan to Share IPD: No